CLINICAL TRIAL: NCT07102628
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate Efficacy and Safety of Early in Hospital Initiation of Inclisiran Treatment in Patients With Acute Coronary Syndromes: Victorion - RIDES
Brief Title: Evaluation of Efficacy and Safety of Early in Hospital Initiation of Inclisiran Treatment in Patients With Acute Coronary Syndromes
Acronym: ACS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CKJX839A12309; 2025-521670-34 (EudraCT Number)
Record Dates: First submitted 2025-07-31; First posted 2025-08-04 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Acute Coronary Syndrome
Keywords: KJX839; Acute Coronary Syndrome; ACS; NSTEMI; STEMI; Inclisiran; LDL-C; Hyperlipidemia
MeSH Terms: conditions — Acute Coronary Syndrome; Non-ST Elevated Myocardial Infarction; ST Elevation Myocardial Infarction; Hyperlipidemias | interventions — ALN-PCS

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inclisiran sodium 300 mg s.c. + Standard treatment (Experimental): * Inclisiran sodium 300 mg subcutaneous (s.c.) on top of HIS (+/- LLT) or non-statin LLT in statin intolerant participants
  * KJX839 284 mg / 1.5 mL (Dose: 300 mg)
  * Pharmaceutical Dosage Form: solution for subcutaneous injection
  Interventions: Drug: Inclisiran
- Matching placebo + Standard treatment (Placebo Comparator): * Matching placebo on top of HIS (+/- LLT) or non-statin LLT in statin intolerant participants
  * KJX839 Placebo / 1.5 mL (Dose: 0 mg)
  * Pharmaceutical Dosage Form: solution for subcutaneous injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — The participants will receive placebo subcutaneous at randomization (Day 1, Baseline visit) and Day 90
  Arms: Matching placebo + Standard treatment
Drug: Inclisiran — The participants will receive Inclisiran sodium 300 mg subcutaneous at randomization (Day 1, Baseline visit) and Day 90
  Arms: Inclisiran sodium 300 mg s.c. + Standard treatment

SUMMARY:
The purpose of this trial is to learn about the effects of inclisiran in people with serious heart conditions (acute coronary syndromes), when this treatment is started early after hospital admission. To do this, researchers will test the effects of inclisiran compared to placebo, when given with standard treatment.

DETAILED DESCRIPTION:
This is a multicenter, prospective, randomized, double-blind, placebo-controlled, two arms, parallel groups clinical trial in participants experiencing an ACS (STEMI or NSTEMI) of recent onset. The study drug treatment (inclisiran/placebo) will be initiated at randomization (Day 1) and before discharge.

The study consists of:

1. Screening visit within 7 days (≤ 7 days) from hospital admission. Screening visit might happen at hospital admission day or any time after hospital admission and before randomization (Day 1).
2. Randomization/Baseline visit (Day 1) within 7 days (≤ 7 days) from hospital admission and before or at day of discharge.

   The discharge can happen any time after randomization and first study drug administration (Day 1).
3. Double-blinded treatment period (150 days).
4. Scheduled safety calls in between visits during the double-blind treatment period (they do not replace on-site visits)
5. Safety Follow-up call (30 days after EOS visit)

Screening and randomization visits must happen during the in-hospital phase, within 7 days (≤ 7 days), and before discharge. The Screening period, of no more than 6 days after the date of hospital admission, will be used to determine if patients qualify to enter the double-blind treatment phase of the study. Screening and Randomization/Day 1 visits cannot occur on the same day. The overall study duration is 150 days.

ELIGIBILITY:
Inclusion Criteria:

Participant eligible for inclusion in this study must meet all the following criteria:

At Screening:

1. Signed informed consent must be obtained prior to participation in the study.
2. Males and females, ≥18 years of age at the time of providing written informed consent.
3. Ability to understand study's requirements and provide informed consent and comply with all required study procedures.
4. Hospitalization for a ACS event (STEMI or NSTEMI).
5. Receiving treatment for the qualifying ACS event, according to clinical judgement, by means of medical treatment alone or percutaneous coronary revascularization.
6. Had a successful PCI (with or without stent) for the qualifying event if a PCI was required.
7. LDL-C value at the Screening visit measured by the local lab of:

   * LDL-C ≥70 mg/dL in participant previously treated with high-intensity statin (atorvastatin ≥40 mg/day or rosuvastatin ≥20 mg/day) or equivalent as per national guidelines and local regulation for at least 4 weeks before screening or
   * LDL-C ≥100 mg/dL in participant previously treated with low/moderate-intensity statin for at least 4 weeks before screening or
   * LDL-C ≥125 mg/dL in participant previously not treated with statins for at least 4 weeks before screening, or who never received statins (including statin intolerant participants).

   At Randomization:
8. The participant must have a Baseline fasting LDL-C ≥70 mg/dL (local lab assessment) to be eligible for randomization.
9. Randomization within 7 days (≤ 7 days) following hospital admission for the qualifying ACS event and before/at discharge.

Exclusion Criteria:

Participant meeting any of the following criteria is not eligible for inclusion in this study.

Only for Japan: For exclusion criteria 6, investigator judgment should be documented in the source data document.

1. Participant who is clinically unstable during hospitalization for the qualifying ACS event, defined by any of the following events within 24 hours prior to randomization:

   * Hemodynamic instability: hypotension, defined as sustained systolic blood pressure of <90 mmHg due to cardiac failure with associated symptoms requiring inotropes
   * Arrhythmic events: Ventricular storm (e.g., torsade, ventricular tachycardia, ventricular flutter)
   * Cardiogenic shock or mechanical complication of myocardial infarction
   * New York Heart Association (NYHA) class IV heart failure
   * Left ventricular ejection fraction <20% at randomization (after all treatment procedures, based on the latest assessment of the LVEF using invasive or non-invasive assessment modalities)
   * Uncontrolled severe hypertension: systolic blood pressure >180 mmHg or diastolic blood pressure >110 mmHg prior to randomization despite antihypertensive therapy.
2. Participant who has undergone or is scheduled to undergo CABG for treatment of the qualifying ACS event.
3. Active liver disease defined as: (i) any known current infectious, neoplastic, or metabolic pathology of the liver or (ii) alanine aminotransferase (ALT) elevation >3x ULN or aspartate aminotransferase (AST) elevation >3x ULN, or total bilirubin elevation >2x ULN (except participant with Gilbert's syndrome) at the Screening visit, in the context of an ACS, and assessed as related to the index event and/or treatment procedures (such as PCI). Eligibility will be based on Investigator's judgement for participant who will be randomized.
4. Renal insufficiency (eGFR <30 mL/min/1.73m2) at the Screening visit.
5. Fasting triglycerides value >400 mg/dL (4.52 mmol/L; assessed by local labs) at randomization visit.
6. Participant, who based on the Investigator's judgement, could reach the LDL-C target value of <55 mg/dL after 4 weeks on statin treatment only.
7. Secondary hypercholesterolemia (based on medical history).
8. Homozygous familial hypercholesterolemia (based on medical history).
9. Participant on apheresis at the Screening visit.
10. Ongoing or medical history of myopathy at the Screening visit.
11. CK values ≥5x ULN at Screening visit and confirmed by repeat test during Screening (local lab) , in the context of an ACS, and assessed as related to the index event and/or treatment procedures (such as PCI) eligibility will be based on Investigator's judgement for participant who will be randomized (who will be switched to or initiated on the protocol-specified dose of high-intensity statin of atorvastatin ≥40 mg QD or rosuvastatin ≥20 mg QD). Unless a more stringent CK value threshold is mandated by a local regulatory authority (e.g., ≥3x ULN in Korea according to MFDS internal guideline).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-10-03 (Actual); Primary Completion 2027-02-15 (Estimated); Study Completion 2027-02-15 (Estimated)

PRIMARY OUTCOMES:
Percent change in LDL-C | From baseline to Day 150
  To demonstrate the superiority of inclisiran treatment compared to placebo, when initiated before/at discharge, in combination with standard of care (SoC) (statin therapy +/- LLT (Lipid Lowering Therapy) or non-statin treatment in case of documented statin intolerance) on LDL-C reduction at Day 150

SECONDARY OUTCOMES:
Participants achieving LDL-C <70 mg/dL (yes, no) | At Day 150
  To assess the proportion of participants reaching pre-specified LDL-C target (<70 mg/dL) on inclisiran treatment compared to placebo, on top of SoC at Day 150
Participants achieving LDL-C <55 mg/dL (yes, no) | At Day 150
  To assess the proportion of participants reaching pre-specified LDL-C target (<55 mg/dL) on inclisiran treatment compared to placebo, on top of SoC at Day 150
Participants achieving LDL-C <100 mg/dL (yes, no) (among the subset of participants with LDL-C ≥100 mg/dL at baseline) | At Day 150
  To assess the proportion of participants reaching pre-specified LDL-C target (<100 mg/dL) on inclisiran treatment compared to placebo, on top of SoC at Day 150
Participants achieving ≥50% reduction from baseline in LDL-C (yes, no) | At Day 150
  To assess the proportion of participants reaching pre-specified LDL-C target (≥50% reduction from baseline) on inclisiran treatment compared to placebo, on top of SoC at Day 150
Percent change from baseline to mean LDL-C over the double-blind treatment period (averaged over all post-baseline visits) | From baseline to Day 30, Day 90 and Day 150
  To assess the mean change (averaged over all post-baseline visits), and the change by visit, from baseline in LDL-C for participants receiving inclisiran treatment compared to placebo, on top of SoC
Absolute change from baseline to mean LDL-C over the double-blind treatment period (averaged over all post-baseline visits) | From baseline to Day 30, Day 90 and Day 150
  To assess the mean change (averaged over all post-baseline visits), and the change by visit, from baseline in LDL-C for participants receiving inclisiran treatment compared to placebo, on top of SoC
Percent change in LDL-C | From baseline to Day 30 and Day 90
  To assess the mean change (averaged over all post-baseline visits), and the change by visit, from baseline in LDL-C for participants receiving inclisiran treatment compared to placebo, on top of SoC
Absolute change in LDL-C | From baseline to Day 30, Day 90 and Day 150
  To assess the mean change (averaged over all post-baseline visits), and the change by visit, from baseline in LDL-C for participants receiving inclisiran treatment compared to placebo, on top of SoC
Percent change and absolute change in PCSK9 | From baseline to Day 30, Day 90 and Day 150
  To assess the change of PCSK9 from baseline to Day 150 in participants on inclisiran treatment compared to placebo, on top of SoC
Percent change and absolute change from baseline in: apoB, VLDL, non-HDLC, HDL-C, total cholesterol and triglycerides | At Day 150
  To assess the change in plasma lipoproteins and triglycerides from baseline to Day 150 in participants on inclisiran treatment compared to placebo, on top of SoC

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (14):
- China (3):
  - Novartis Investigative Site, Luoyang, Henan
  - Novartis Investigative Site, Wenzhou, Zhejiang
  - Novartis Investigative Site, Shanghai
- Novartis Investigative Site, Hong Kong, Hong Kong, Hong Kong
- Japan (5):
  - Novartis Investigative Site, Chikushino-shi, Fukuka
  - Novartis Investigative Site, Kitakyushu, Fukuoka
  - Novartis Investigative Site, Kamakura, Kanagawa
  - Novartis Investigative Site, Sagamihara, Kanagawa
  - Novartis Investigative Site, Bunkyo Ku, Tokyo
- South Korea (2):
  - Novartis Investigative Site, Seoul, Seoul
  - Novartis Investigative Site, Seoul
- Switzerland (3):
  - Novartis Investigative Site, Bern
  - Novartis Investigative Site, Geneva
  - Novartis Investigative Site, Lucerne

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com